CLINICAL TRIAL: NCT06420830
Title: Title Valve Performance of the SAPIEN 3 Ultra RESILIA Valve: a Prospective Registry with Central Echocardiography Analysis.
Brief Title: Valve Performance of the SAPIEN 3 Ultra RESILIA Valve: a Prospective Registry with Central Echocardiography Analysis.
Status: Recruiting | Type: Observational
Sponsor: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Responsible Party: Principal Investigator, Josep Rodes-Cabau, Principal Investigator, Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Other Study IDs: RESILIA
Record Dates: First submitted 2024-05-15; First posted 2024-05-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-05

CONDITIONS: Aortic Valve Stenosis; Transcatheter Aortic Valve Replacement
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: SAPIEN 3 Ultra RESILIA Valve — Patients with severe aortic stenosis undergoing transarterial TAVR with the SAPIEN 3 Ultra RESILIA valve.

SUMMARY:
The issue of valve durability has become one of the most important aspects in the TAVR field in recent years since transcatheter aortic valve replacement has been progressively applied to younger patients with a low co-morbidity burden. The SAPIEN 3 Ultra RESILIA valve represents the last generation of the SAPIEN valve system and includes several important iterations (newer leaflet calcium-blocking technology targeting calcium-attracting free aldehydes, dry tissue storage, newer skirt textile design) that should translate into a favorable impact on valve durability at mid- to long- term follow-up

DETAILED DESCRIPTION:
Prospective observational registry including patients with severe aortic stenosis undergoing TAVR with the SAPIEN 3 Ultra RESILIA valve. All patients who will survive the procedure will undergo a clinical and echocardiographic follow-up at 1-3 months (± 15 days), at 1-year (±30 days), 3-5 year (±30 days), 6-8 year (±30 days) and 9-10 year (±30 days) after valve implantation. Transthoracic echocardiography (TTE) exams (baseline, 1-3-month, 1 year, 3-5 years, 6-8 years, and 9-10 years post-procedure) will be evaluated in a Centralized Echocardiographic Core Lab at the Quebec Heart and Lung Institute. The measurements obtained in the Core Lab regarding transvalvular gradient, EOA, PPM and PVL at 1-3 months will determine the primary outcome of the study.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria - Patients with severe aortic stenosis undergoing transarterial TAVR with the SAPIEN 3 Ultra RESILIA valve.
* Successful valve implantation of the SAPIEN 3 Ultra RESILIA valve.

VARC-3- defined technical success defined as:

* Freedom from mortality
* Successful access, delivery of the device, and retrieval of the delivery system
* Correct positioning of a single prosthetic heart valve into the proper anatomical location
* Freedom from surgery or intervention related to the device (excluding permanent pacemaker) or to a major vascular or access related, or cardiac structural complication - Absence of severe procedural or in-hospital complications (VARC-3 definitions): mortality, stroke, bleeding type 2-4, myocardial infarction, need for a second valve, valve embolization, coronary obstruction, annular rupture.

Exclusion Criteria:

* Age >80 years
* Severe pulmonary disease (FEV1 <50% predicted or need for home oxygen)
* Severe renal dysfunction (eGFR <30 ml/min/1.73m2)
* Frailty (Clinical Frailty Scale > 4)
* Severe coronary disease (SYNTAX score >32)
* Left ventricular ejection fraction ≤30%
* Moderate-to-severe mitral regurgitation
* Severe tricuspid regurgitation
* Pulmonary systolic pressure >60 mmHg
* STS-PROM >5%
* Any disease leading to a life expectancy <5 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population Patients with severe aortic stenosis undergoing transcatheter aortic valve replacement (TAVR) with the SAPIEN 3 Ultra RESILIA valve.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2034-09-01 (Estimated)

PRIMARY OUTCOMES:
Transvalvular gradient | 1-3 months
  Residual (peak and mean) transvalvular gradient
Effective orifice area (EOA) | 1-3 months
  EOA evaluated by echocardiography imaging
Prosthesis-patient mismatch | 1-3 months
  Moderate or severe prothesis-patient mismatch (defines as an index aortic valve area 0.85-0.66 cm2/m2 (moderate), ≤0.65 cm2/m2 (severe) for patient with BMI ˂30km/m2 and 0.70-0.56 cm2/m2 (moderate), ≤0.55 cm2/m2 (severe) for patient with BMI ≥30km/m2 and/or moderate-severe aortic regurgitation (AR) (VARC-3 definition).
Paravalvular leaks | 1-3 months
  Paravalvular leaks evaluated by echocardiography imaging

SECONDARY OUTCOMES:
Transvalvular gradient | 1-, 3-5-, 6-8-, and 9-10-year follow-up.
  Residual (maximal and mean) transvalvular gradient
Effective orifice area (EOA) | 1-, 3-5-, 6-8-, and 9-10-year follow-up.
  EOA evaluated by echocardiography imaging
Bioprosthetic valve dysfunction | 1-, 3-5-, 6-8-, and 9-10-year follow-up.
  Bioprosthetic valve dysfunction evaluated by VARC3 criteria
Paravalvular leaks | 1-, 3-5-, 6-8-, and 9-10-year follow-up.
  Paravalvular leaks evaluated by echocardiography imaging
Bioprosthetic valve dysfunction | yearly
  Incidence rate (per 100 patient-years) of bioprosthetic valve dysfunction (stage 2 or 3)
Bioprosthetic valve failure | yearly
  Incidence rate (per 100 patient-years) of bioprosthetic valve failure
Bioprosthetic valve failure | 1-, 3-5-, 6-8-, and 9-10-year follow-up.
  Bioprosthetic valve failure evaluated by VARC3 criteria
Clinical events | 1month and yearly up to 10-year
  Individual: mortality, stroke, bleeding type 2-4, cardiac rehospitalization, heart failure rehospitalization
Valve thrombosis | 1-3 months and yearly up to 10-year
  Number of patients with valve thrombosis
Valve endocarditis | 1-3 months and yearly up to 10-year
  Number of patients with valve endocarditis

CONTACTS AND LOCATIONS:
Overall Officials: Josep Rodés-Cabau, MD, Principal Investigator — IUCPQ-UL; Emilie Pelletier beaumont, MSc, Study Director — Fondation IUCPQ
Locations (1):
- IUCPQ, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Writing Committee Members; Otto CM, Nishimura RA, Bonow RO, Carabello BA, Erwin JP 3rd, Gentile F, Jneid H, Krieger EV, Mack M, McLeod C, O'Gara PT, Rigolin VH, Sundt TM 3rd, Thompson A, Toly C; ACC/AHA Joint Committee Members; O'Gara PT, Beckman JA, Levine GN, Al-Khatib SM, Armbruster A, Birtcher KK, Ciggaroa J, Deswal A, Dixon DL, Fleisher LA, de las Fuentes L, Gentile F, Goldberger ZD, Gorenek B, Haynes N, Hernandez AF, Hlatky MA, Joglar JA, Jones WS, Marine JE, Mark D, Palaniappan L, Piano MR, Spatz ES, Tamis-Holland J, Wijeysundera DN, Woo YJ. 2020 ACC/AHA guideline for the management of patients with valvular heart disease: A report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. J Thorac Cardiovasc Surg. 2021 Aug;162(2):e183-e353. doi: 10.1016/j.jtcvs.2021.04.002. Epub 2021 May 8. No abstract available. PMID 33972115
- [Background] Vahanian A, Beyersdorf F, Praz F, Milojevic M, Baldus S, Bauersachs J, Capodanno D, Conradi L, De Bonis M, De Paulis R, Delgado V, Freemantle N, Gilard M, Haugaa KH, Jeppsson A, Juni P, Pierard L, Prendergast BD, Sadaba JR, Tribouilloy C, Wojakowski W; ESC/EACTS Scientific Document Group. 2021 ESC/EACTS Guidelines for the management of valvular heart disease. Eur Heart J. 2022 Feb 12;43(7):561-632. doi: 10.1093/eurheartj/ehab395. No abstract available. PMID 34453165
- [Background] Mack MJ, Leon MB, Thourani VH, Makkar R, Kodali SK, Russo M, Kapadia SR, Malaisrie SC, Cohen DJ, Pibarot P, Leipsic J, Hahn RT, Blanke P, Williams MR, McCabe JM, Brown DL, Babaliaros V, Goldman S, Szeto WY, Genereux P, Pershad A, Pocock SJ, Alu MC, Webb JG, Smith CR; PARTNER 3 Investigators. Transcatheter Aortic-Valve Replacement with a Balloon-Expandable Valve in Low-Risk Patients. N Engl J Med. 2019 May 2;380(18):1695-1705. doi: 10.1056/NEJMoa1814052. Epub 2019 Mar 16. PMID 30883058
- [Background] Popma JJ, Deeb GM, Yakubov SJ, Mumtaz M, Gada H, O'Hair D, Bajwa T, Heiser JC, Merhi W, Kleiman NS, Askew J, Sorajja P, Rovin J, Chetcuti SJ, Adams DH, Teirstein PS, Zorn GL 3rd, Forrest JK, Tchetche D, Resar J, Walton A, Piazza N, Ramlawi B, Robinson N, Petrossian G, Gleason TG, Oh JK, Boulware MJ, Qiao H, Mugglin AS, Reardon MJ; Evolut Low Risk Trial Investigators. Transcatheter Aortic-Valve Replacement with a Self-Expanding Valve in Low-Risk Patients. N Engl J Med. 2019 May 2;380(18):1706-1715. doi: 10.1056/NEJMoa1816885. Epub 2019 Mar 16. PMID 30883053
- [Background] Montarello NJ, Willemen Y, Tirado-Conte G, Travieso A, Bieliauskas G, Sondergaard L, De Backer O. Transcatheter aortic valve durability: a contemporary clinical review. Front Cardiovasc Med. 2023 May 9;10:1195397. doi: 10.3389/fcvm.2023.1195397. eCollection 2023. PMID 37229228
- [Background] Ferreira-Neto AN, Rodriguez-Gabella T, Guimaraes L, Freitas-Ferraz A, Bernier M, Figueiredo Guimaraes C, Pasian S, Paradis JM, Delarochelliere R, Dumont E, Mohammadi S, Kalavrouziotis D, Cote M, Pibarot P, Rodes-Cabau J. Multimodality evaluation of transcatheter structural valve degeneration at long-term follow-up. Rev Esp Cardiol (Engl Ed). 2021 Mar;74(3):247-256. doi: 10.1016/j.rec.2020.02.002. Epub 2020 Apr 8. English, Spanish. PMID 32278660
- [Background] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243